CLINICAL TRIAL: NCT06270771
Title: OURA Ring Wearable Testing in MDS Patients: a Feasibility and Discovery Pilot Study
Acronym: OURA MDS
Status: Recruiting | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 5823
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: MDS; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; RARS-T
Keywords: transfusion dependent; transfusion independent; OURA ring
MeSH Terms: conditions — Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfusion Dependent: Patients who are currently receiving transfusions will be assigned to this cohort
  Interventions: Device: OURA Ring
- Transfusion Independent: Patients who are not currently receiving transfusions will be assigned to this cohort
  Interventions: Device: OURA Ring

INTERVENTIONS:
Device: OURA Ring — The OURA ring (https://ouraring.com) is a light-weight wearable device in the form of a ring that has several microsensors enabling detection of heart rate, blood oxygen level, skin temperature, and movement. The OURA ring and application can synthesize the sensory data to generate physiologic information such as sleep, activity level, resting heart rate, heart rate variability, respiratory rate, and more. The OURA ring is water resistant and has up to 5-7 days of battery life and can be fully charged in 20-80 minutes. It communicates with the OURA app and commonly used Smartphone health apps via Bluetooth connectivity with automatic syncing every week.

SUMMARY:
A prospective, single center, single arm phase 2 cohort feasibility study of the OURA ring in adult MDS patients. Patients with MDS will wear the OURA ring and upload biometrics weekly. Quality of life measures will be clinically evaluated and correlated with biometrics. We hypothesize that it will be feasible for MDS patients to wear the OURA ring 70% of the time for 3 months.

DETAILED DESCRIPTION:
This is a single-centre feasibility study involving two groups of patients (transfusion-dependent MDS and non-transfusion dependent MDS), each enrolling 30 patients. Eligible patients who consent to the study will be provided with the OURA ring sizing kit to determine their ring size. Baseline characteristics will be collected, including the following information if available:

* Patient demographics such as age, sex, history of cancer
* MDS disease characteristics: date of diagnosis, IPSS and IPSS-R score, transfusion status, transfusion schedule, MDS specific treatment and concomittent medications
* Laboratory data: hemoglobin, MCV, RDW, WBC, reticulocyte count, creatinine clearance, bilirubin, ALT, AST, LDH, ferritin

The correctly sized OURA ring will be ordered and provided to the patient within 4 weeks during their Baseline visit at "week 0". At this time, technological assistance will be provided for correctly wearing the ring, installation of the OURA app to their smartphone, and teaching the patient how to sync the OURA ring to their device. During this visit, patients will have their first clinical assessment which includes a physical exam, vitals, height and weight, as well as the 4-metre walk test and the administration of the study questionnaires (ECOG score, clinical frailty score, QLQ-C30, QUALMS, EQ-5D, global fatigue scale, and the Lawton-Brody instrumental activity of daily living (IADL) scale.

Patients will be given study forms to take home and complete based on the schedule listed in Appendix A. This includes a daily log of their global fatigue score, and a section for descriptive annotation of significant events in the day. Once every 7 days, patients will fill in the QLQ-C30, PROMIS-fatigue, QUALMS physical functioning subscale and synchronize the OURA ring data onto their smartphone.

Patients will have monthly follow-up appointments at 1 and 2 months into the study. At these times, clinical events in the month will be reviewed, including whether they had transfusions, hospitalizations, or major health events. Patients' OURA ring data will be reviewed. Depending on OURA ring results, the physician involved may determine to order additional investigations or referrals (such as sleep clinic assessment or cardiology referrals).

At month 3, patients will have their study exit visit. Data from the OURA ring app will be downloaded and a debrief will occur to qualitatively gauge the experience of a wearable device.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 or older
4. Able to read, write and speak English or French (non-English or French speaking patients may participate if appropriate translation is used)
5. Diagnosed with Myelodysplastic Syndrome using WHO 2022 criteria (12) all risk groups
6. Ability to wear the OURA ring and operate the associated smart-phone app, and willing to adhere to the study regimen

Exclusion Criteria:

1. Performance status ECOG > 3.
2. Cognitive or physical impairment preventing the usage or utilization of the OURA ring and smart phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 Adult patients with MDS of which 30 are transfusion-dependent and 30 are non-transfusion dependent. There are no limitations with regards to age or gender.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of patients with MDS wearing the OURA ring | 3 months
  Feasibility will be defined as being worn 70% of the time and uploaded to a web-based database weekly x 3 months.

SECONDARY OUTCOMES:
Exploratory correlations between physiologic changes captured by the wearable device and physical functioning | 2 years
  Correlation between self-rated fatigue, physical functioning with steps taken, calories burned/day, sleep, readiness scores; Correlation between resting heart rate, heart rate variability, respiratory rate, oxygen saturation with hemoglobin, transfusion dependence, dates of transfusion, and unplanned healthcare encounters

CONTACTS AND LOCATIONS:
Locations (1):
- Sunnybrook Health Sciences Research Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No